CLINICAL TRIAL: NCT03006679
Title: A Phase IIIb, Multicenter, Double-Blind, Randomized, Comparative Study to Evaluate the Efficacy, Safety, and Tolerability of Meropenem-Vaborbactam Versus Piperacillin/Tazobactam in the Treatment of Hospital-Acquired Bacterial Pneumonia and Ventilator-Associated Bacterial Pneumonia in Hospitalized Adults (TANGO III)
Brief Title: A Study of Meropenem-Vaborbactam Versus Piperacillin/Tazobactam in Participants With Hospital-Acquired and Ventilator-Associated Bacterial Pneumonia
Acronym: TANGOIII
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Rempex 509
Record Dates: First submitted 2016-12-15; First posted 2016-12-30 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Hospital-Acquired Bacterial Pneumonia; Ventilator-Associated Bacterial Pneumonia; Hospital-Acquired Pneumonia; Ventilator-Associated Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated | interventions — meropenem and vaborbactam; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Meropenem-Vaborbactam HABP (Experimental): Participants with a clinical diagnosis of HABP will be treated with meropenem 2 grams (g) and vaborbactam 2 g in 250 milliliters (mL) infused intravenously for 3 hours every 8 hours for 7 days to a maximum of 14 days.
  Interventions: Drug: Meropenem-Vaborbactam
- Piperacillin/Tazobactam HABP (Active Comparator): Participants with a clinical diagnosis of HABP will be treated with piperacillin 4 g and tazobactam 0.5 g in 100 mL infused intravenously for 30 minutes every 6 hours for 7 days to a maximum of 14 days.
  Interventions: Drug: Piperacillin/Tazobactam
- Meropenem-Vaborbactam VABP (Experimental): Participants with a clinical diagnosis of VABP will be treated with meropenem 2 g and vaborbactam 2 g in 250 mL infused intravenously for 3 hours every 8 hours for 7 days to a maximum of 14 days.
  Interventions: Drug: Meropenem-Vaborbactam
- Piperacillin/Tazobactam VABP (Active Comparator): Participants with a clinical diagnosis of VABP will be treated with piperacillin 4 g and tazobactam 0.5 g in 100 mL infused intravenously for 30 minutes every 6 hours for 7 days to a maximum of 14 days.
  Interventions: Drug: Piperacillin/Tazobactam

INTERVENTIONS:
Drug: Meropenem-Vaborbactam — meropenem 2 g and vaborbactam 2 g
  Other Names: Carbavance
  Arms: Meropenem-Vaborbactam HABP; Meropenem-Vaborbactam VABP
Drug: Piperacillin/Tazobactam — piperacillin 4 g and tazobactam 0.5 g
  Other Names: Zosyn
  Arms: Piperacillin/Tazobactam HABP; Piperacillin/Tazobactam VABP

SUMMARY:
The purpose of this study is to determine the efficacy, safety, tolerability, and pharmacokinetics (PK) of meropenem-vaborbactam compared to piperacillin/tazobactam for 7 to 14 days in the treatment of hospitalized adults who meet clinical, radiographic, and microbiological criteria for hospital-acquired bacterial pneumonia (HABP) or ventilator-associated bacterial pneumonia (VABP).

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to comply with all study procedures and provide a signed written informed consent prior to any study-specific procedures; however, if unable to do so, the participant's legally authorized representative may provide written consent as approved by institutional-specific guidelines. Participants who are unconscious or considered by the investigator to be clinically unable to consent at Screening and who are entered into the study by the consent of a legally authorized representative, should provide their own written informed consent for continuing to participate in the study as soon as possible on recovery, as applicable in accordance with local regulations.
2. Hospitalized male or female participants, ≥18 years of age.
3. Females must be surgically sterile or at least 2 years postmenopausal, or if of childbearing potential, have a negative screening urine pregnancy test and be willing to practice sexual abstinence or use an accepted form of contraception with her partner (for example, barrier or hormonal methods) during treatment and for at least 28 days after the last dose of study drug.
4. Expectation, in the opinion of the Investigator, that the participant's infection will require treatment with IV antibiotics for a minimum of 7 days.
5. Have a confirmed diagnosis of HABP or VABP requiring antibiotic therapy by meeting all clinical, microbiological, and radiographic criteria as defined in the following:

For HABP participants:

To meet the study definition of HABP, participants must meet all of the following clinical, microbiological, and radiographic criteria:

1. A chest radiograph (chest X-ray [CXR], magnetic resonance imaging [MRI] or computed tomography [CT]) reveals the presence of new or progressive pulmonary infiltrate(s) consistent with bacterial pneumonia within 48 hours prior to randomization.
2. Onset of symptoms at least 48 hours after hospitalization or within 7 days after discharge from an inpatient acute or chronic care facility (for example, long-term care, rehabilitation center, hospital, or skilled nursing home).
3. Have at least one of the following:

   1. Temperature ≥38.0 degrees Celsius (100.4 degrees Fahrenheit) or ≤35 degrees Celsius (95.0 degrees Fahrenheit).
   2. Peripheral white blood cell (WBC) count ≥10,000 cells/cubic millimeter (mm^3) or ≤4,500 cells/mm^3.
   3. ≥15 percent immature neutrophils (band forms) regardless of total WBC count.
4. Have at least one of the following:

   1. New onset of cough or expectorated sputum production (or worsening of baseline cough).
   2. Auscultatory findings on pulmonary examination consistent with bacterial pneumonia or pulmonary consolidation (for example, rales, dullness on percussion, bronchial breath sounds, or ego phony).
   3. Dyspnea or tachypnea (that is, respiratory rate greater than 25 breaths/minute).
   4. Hypoxemia (O2 saturation ≤90 percent or pO2 ≤60 millimeters of mercury [mmHg] while breathing room air, or worsening of the O2 saturation/FiO2).
   5. New onset need for mechanical ventilation.
   6. A deep respiratory secretion specimen that was collected within 48 hours prior to randomization and after development of clinical signs and symptoms of HABP (ideally prior to administration of systemic antimicrobial therapy). This can be obtained via a sputum sample (expectorated sputum), bronchoalveolar lavage (BAL) (including protected BAL or mini-BAL), protected specimen brush (PSB), endotracheal tube aspirate (ETA), pleural fluid, or lung parenchyma (open-lung, transthoracic, or transbronchial biopsy).
   7. This deep respiratory secretion sample must meet adequacy criteria for testing, and be sent to the local or regional laboratory for Gram stain and culture (results of Gram stain and culture do not have to be available for enrollment).

For VABP participants:

To meet the study definition of VABP, participants must meet all of the following clinical, microbiological, and radiographic criteria:

1. A chest radiograph (CXR, MRI or CT) revealing the presence of new or progressive pulmonary infiltrate(s) consistent with bacterial pneumonia within 48 hours prior to randomization.
2. Receiving mechanical ventilation via endotracheal intubation or tracheostomy for greater than or equal to 48 hours.
3. Have at least one of the following:

   1. Temperature ≥38.0 degrees Celsius (100.4 degrees Fahrenheit) or ≤35 degrees Celsius (95.0 degrees Fahrenheit).
   2. Peripheral white blood cell (WBC) count ≥10,000 cells/mm^3 or ≤4,500 cells/mm^3.
   3. ≥15 percent immature neutrophils (band forms) regardless of total WBC count.
4. Have at least one of the following:

   1. New onset of purulent respiratory secretions from the lungs or new onset of or increased need for respiratory secretion suctioning.
   2. Auscultatory findings on pulmonary examination consistent with bacterial pneumonia or pulmonary consolidation (for example, rales, dullness on percussion, bronchial breath sounds, or egophony).
   3. Worsening gas exchange (ratio of partial pressure of arterial oxygen to fraction of inspired oxygen [PaO2/FiO2] ≤240 or PaO2 ≤60 mmHg) leading to acute changes to the ventilator support system (minimum daily FiO2 values increased by at least 0.20 over the daily minimum FiO2 in the preceding 48 hours, or minimum daily positive end- expiratory pressure (PEEP) values increased by at least 3 centimeters (cm) H2O over the daily minimum PEEP in the preceding 48 hours).
5. A deep respiratory secretion specimen must be collected within 48 hours prior to randomization and after development of clinical signs and symptoms of VABP (ideally prior to administration of systemic antimicrobial therapy). This can be obtained via BAL (including protected BAL or mini-BAL), PSB, or ETA, pleural fluid, or lung parenchyma (open-lung, transthoracic, or transbronchial biopsy).
6. The above deep respiratory secretion sample must meet adequacy criteria for testing and be sent to the local or regional laboratory for Gram stain and culture (results of Gram stain and culture do not have to be available for enrollment).

Exclusion Criteria:

Participants who meet any of the following exclusion criteria will not be enrolled in the study:

1. History of any severe hypersensitivity to any beta-lactam antibiotic (for example, cephalosporins, penicillins, or carbapenems).
2. History of any severe allergic reaction that would preclude the use of either all aminoglycosides or adjunctive gram-positive antimicrobials (that is, allergy to both glycopeptides and oxazolidinones).
3. Requirement or anticipated need for additional systemic antibiotic (other than study drug) or antifungal, including prophylactic antimicrobials and antifungals.
4. Requirement or anticipated need for more than 14 days of systemic antimicrobial therapy to treat HABP or VABP.
5. Known deep-tissue infection (including undrained abscess, meningitis, endocarditis, or osteomyelitis) within 7 days prior to randomization.
6. Participant has received more than 24 hours of any potentially effective systemic antibacterial therapy for the current episode of HABP or VABP within 72 hours before randomization. Exceptions:

   1. Evidence of clinical failure of the current episode of HABP or VABP (for example, worsening signs and symptoms) following at least 48 hours of prior systemic antimicrobial therapy (participants with evidence of clinical failure of piperacillin/tazobactam are not eligible for inclusion), or
   2. The clinical symptoms and signs of the current episode of HABP or VABP started at least 48 hours after the prior antibacterial therapy was initiated.
7. Pulmonary disease that precludes evaluation of a therapeutic response (including, but not limited to, lung cancer, active tuberculosis, cystic fibrosis, granulomatous disease, fungal pulmonary infection, pulmonary embolism, lung abscess, pleural empyema, or post obstructive pneumonia).
8. Known human immunodeficiency virus (HIV) positivity and meets an acquired immune deficiency syndrome (AIDS)-defining illness or has a documented CD4 count <200/ microliter (μL) within the past year.
9. Treatment within 30 days prior to enrollment with bone-marrow suppressive chemotherapy (non-bone marrow suppressive chemotherapy is permitted), high dose steroids, immunosuppressive medications for transplantation, or medications for rejection of transplantation.
10. Fulminant hepatitis; current cirrhosis or clinical manifestations of end-stage liver disease (for example, ascites or hepatic encephalopathy); acute hepatic failure or acute decompensation of chronic hepatic failure; or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level greater than 5-fold the upper limit of normal or total bilirubin greater than 3-fold the upper limit of normal using local or regional laboratory reference values.
11. Requirement for peritoneal dialysis or continuous renal replacement therapy (including continuous venovenous hemofiltration [CVVH], continuous venovenous hemodialysis [CVVHD], and continuous venovenous hemodiafiltration [CVVHDF]) (Note, standard intermittent hemodialysis is not exclusionary).
12. Females who are pregnant or breastfeeding.
13. Participation in any study involving administration of an investigational agent or device within 30 days prior to randomization into this study or previous participation in the current study or any study of vaborbactam or meropenem vaborbactam.
14. Any condition that would make the participant, in the opinion of the Investigator, unsuitable for the study (for example, would place a participant at risk or compromise the quality of the data), including participants with a high likelihood of death within 72 hours after randomization despite adequate antimicrobial therapy for HABP or VABP or participants with a "do not resuscitate" order.
15. An employee of the Investigator or study center with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, or a family member of the employee or the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Participants with All-Cause Mortality at Day 28 in the Intent-to-Treat (ITT) Population | Day 28
Percentage of Participants who Achieve a Clinical Outcome of Cure at the Test of Cure (TOC) Visit in the ITT and Clinically Evaluable (CE) Populations | 12-23 days (TOC visit) after first dose of study drug

SECONDARY OUTCOMES:
Rate of Participants with All-Cause Mortality at Day 14 in the ITT, microbiological Modified ITT (mMITT), CE, and Microbiologically Evaluable (ME) Populations | Day 14
Rate of Participants with All-Cause Mortality at Day 28 in the mMITT, CE, and ME Populations | Day 28
Percentage of Participants with Clinical Outcome of Cure at EOT, TOC, and Last Follow Up (LFU) Visits in the ITT, CE, and ME Populations | 1 day (EOT visit), 12-23 days (TOC visit), and 19-30 days (LFU visit) after first dose of study drug
Percentage of Participants with Clinical Outcome of Cure per Pathogen at EOT, TOC, and LFU Visits in the mMITT and ME Populations | 1 day (EOT visit), 12-23 days (TOC visit), and 19-30 days (LFU visit) after first dose of study drug
Percentage of Participants with Microbiological Eradication Per-Participant and Per-Pathogen Microbiological Response at EOT and TOC visits in the mMITT and ME Populations | 1 day (EOT visit) and 12-23 days (TOC visit) after first dose of study drug
Percentage of Participants who Survive and Did Not Have a "Major Nonfatal Event" (Treatment-Emergent Events of Acute Respiratory Distress Syndrome, Septic Shock, or Pleural Empyema) up to Day 28 in the ITT and CE Populations | Up to Day 28
Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of Meropenem | Days 1 and 3
Pharmacokinetics: Maximum Plasma Concentration (Cmax) of Meropenem | Days 1 and 3
Pharmacokinetics: Time to Maximum Plasma Concentration (Tmax) of Meropenem | Days 1 and 3
Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of Vaborbactam | Days 1 and 3
Pharmacokinetics: Maximum Plasma Concentration (Cmax) of Vaborbactam | Days 1 and 3
Pharmacokinetics: Time to Maximum Plasma Concentration (Tmax) of Vaborbactam | Days 1 and 3